CLINICAL TRIAL: NCT00982371
Title: A Cross-sectional Comparison of Bone Micro-architecture in Postmenopausal Women With Type 2 Diabetes and Age-matched Controls
Brief Title: An Investigation Into Bone Micro-architecture in Women With Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); McMaster University (Other)
Responsible Party: Sponsor
Organization: McMaster University (Other)
Other Study IDs: REB 08-281
Record Dates: First submitted 2009-09-21; First posted 2009-09-23 (Estimated); Last update posted 2012-06-19 (Estimated); Status verified 2012-06

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: type 2 diabetes mellitus; osteoporosis; bone quality; magnetic resonance imaging; fracture; postmenopausal women >65 years old
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Osteoporosis; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Controls: female; >65 years old; BMI >25kg/m2; postmenopausal >5 yrs; NO clinical diagnosis of type 2 diabetes for >5 years (according to Canadian Diabetes Association criteria)
- Type 2 Diabetes: female; >65 years old; BMI >25kg/m2; postmenopausal >5 yrs; clinical diagnosis of type 2 diabetes for >5 years (according to Canadian Diabetes Association criteria)

SUMMARY:
The number of people with type 2 diabetes is growing. This puts a lot of pressure on the health care systems. Type 2 diabetes is often associated with health problems, like poor eyesight, muscle coordination, muscle strength, and blood flow. Poor bone health may also be a concern for people with type 2 diabetes.

A large proportion of people with type 2 diabetes will break a bone in their lifetime. The risk of this happening in older people with type 2 diabetes is greater than the risk in older people without diabetes. Fracturing a bone can be very painful, and lead to serious consequences, especially if the individual experiences a hip fracture. The elevated fracture risk, seen in those with type 2 diabetes, is puzzling because people with type 2 diabetes often appear to have normal, healthy bones compared to people of the same age without diabetes.

Bone micro-structure, which is not assessed by traditional bone densitometry systems (ie: DXA) contributes to overall bone strength.

The hypothesis of this study is that bone micro-structure is of poorer quality (reduced trabecular thickness, increased trabecular spacing) in postmenopausal women with type 2 diabetes, compared to age-matched control participants.

ELIGIBILITY:
Inclusion Criteria:

* female
* >= 65 years old
* postmenopausal for > 5 years (WHO definition of menopause)

Exclusion Criteria:

* currently taking osteoporosis related medication (HRT, SERM, bisphosphonate, PTH, calcitonin, fluoride)
* had cancer in past 10 years, likely to metastasize to bone (ie: breast, lung)
* have intrinsic bone disease (ie: Paget's Disease, Cushings syndrome)
* have untreated malabsorption syndrome (ie: Celiac Disease)
* renal insufficiency (CrCl <30ml/min)
* hyperparathyroidism, hypoparathyroidism
* chronic systemic glucocorticosteroid use > 3mos, dose>2.5mg daily

Min Age: 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: female; >65 years old; BMI >25kg/m2; postmenopausal >5 yrs
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
1 Tesla peripheral MRI assessment at non dominant distal radius: Trabecular bone micro-architecture parameters Tb.Th, Tb.Sp, Tb.N, BV/TV, bone CSA, marrow space | MRI scan complete approximately 1 month after participant is enrolled

SECONDARY OUTCOMES:
Calcium, vitamin D and vitamin K dietary intakes; TUG (sec); grip strength; DXA assessment of hip, lumbar spine, total body; physical activity | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada